CLINICAL TRIAL: NCT04197908
Title: Endoscopic Ultrasound (EUS)-Guided Gallbladder Drainage Instead of Laparoscopic Cholecystectomy for Acute Cholecystitis: A Feasibility Study
Brief Title: EUS-guided Gallbladder Drainage Instead of Laparoscopic Cholecystectomy for Acute Cholecystitis. A Feasibility Study.
Acronym: EGDB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Anthony Teoh, Honorary Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC-2016.609
Record Dates: First submitted 2019-12-06; First posted 2019-12-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Acute Cholecystitis
Keywords: Acute cholecystitis; EUS-guided gallbladder drainage; Laparoscopic cholecystectomy; gallbladder polyp; gallstone
MeSH Terms: conditions — Cholecystitis, Acute; Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUS-guided gallbladder drainage (EGBD) (Experimental): The procedure would be performed with a linear echoendoscope using a 10mm x 10mm or a 15 x 10mm stent. The distal flange of the stent would be deployed under EUS guidance, followed by deployment of the proximal flange under endoscopic guidance. Once deployed, the gallbladder would be completely emptied by suction and irrigation until the effluent through the stent is clean.
  Interventions: Device: EUS-guided gallbladder drainage (EGBD)

INTERVENTIONS:
Device: EUS-guided gallbladder drainage (EGBD) — As listed in the arms description

SUMMARY:
To evaluate the feasibility of performing EGBD as a treatment of acute calculous cholecystitis in patients that are indicated for laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
The gold standard for treatment of acute calculous cholecystitis is laparoscopic cholecystectomy. Recently, gallbladder drainage with EUS-guided gallbladder drainage (EGBD) has been described as a treatment option. However, whether this is an effective treatment option in surgically fit patients are uncertain.

The aim of the current study is to evaluate the feasibility of performing EGBD as a treatment of acute calculous cholecystitis in patients that are indicated for laparoscopic cholecystectomy. The investigators hypothesis that the technique is safe and feasible.

ELIGIBILITY:
Inclusion Criteria:

Consecutive healthy patients aged ≥ 18 years old suffering from acute calculous cholecystitis indicated for laparoscopic cholecystectomy would be included.

Exclusion Criteria:

* Pregnancy
* Patients unwilling to undergo follow-up assessments
* Patients with suspected gangrene or perforation of the gallbladder
* Patients diagnosed with concomitant liver abscess or pancreatitis (defined as elevated serum amylase more than three times the upper limit of normal)
* Patients with duodenal obstruction
* Altered anatomy of the upper gastrointestinal tract due to surgery of the esophagus, stomach and duodenum
* Patients with liver cirrhosis, portal hypertension and/or gastric varices
* Abnormal coagulation: international normalised ratio (INR) > 1.5 and/or platelets < 50.000/mm3
* Previous drainage of the gallbladder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-29 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate | 30 days
  Complete resolution of acute cholecystitis as defined by resolution of fever, pain and change of white cell counts of 10%

SECONDARY OUTCOMES:
Technical success rate | 30 days
  Defined as successful placement of a metal stent between the gallbladder and the duodenum or the stomach
30-day adverse events rate | 30 days
  Adverse events would be graded according to the lexicon of endoscopic adverse events
Stone or polyp recurrences | 3 years
  An ultrasonography of the abdomen would also be arranged yearly to check for recurrence of stones or polyps.
Quality of life scores: Gastrointestinal quality of life index | 3 years
  Gastrointestinal quality of life index
Mortality rate | 3 years
  Death from any cause
Reintervention rate | 3 years
  The number of patients requiring biliary related re-interventions within 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Teoh, Principal Investigator — CUHK
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong, China